CLINICAL TRIAL: NCT01986127
Title: A Randomized, Double-blinded, Placebo-controlled Study on the Effects of Adalimumab Intralesional Intestinal Strictures of Crohn's Disease Patients
Brief Title: Adalimumab Intralesional in Intestinal Strictures of Crohn's Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Sara Varea (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSAI; 2012-001723-12 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-11-18 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Crohn's Disease
Keywords: Crohn disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental): single administration of Adalimumab 80mg diluted in 5ml saline
  Interventions: Drug: Adalimumab
- saline (Placebo Comparator): 5 ml of saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Adalimumab — single intralesional administration during endoscopy process
  Arms: Adalimumab
Drug: placebo — single intralesional administration during endoscopy
  Arms: saline

SUMMARY:
We study if the administration of intralesional Adalimumab (directly injected in the stricture) associated to endoscopic dilatation has a higher success rate at week 8 compared with placebo in patients with Crohn's disease who had confirmed intestinal stenosis (3 stenosis as maximum)

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years
* Patient diagnosed of CROHN´s disease
* Patient with intestinal stenosis length equal or less than 5cm previously confirmed with bowel magnetic resonance imaging (3 stenosis as maximum)
* Stenosis no permeable for endoscopy(12mm in case of accessible stenosis with conventional colonoscopy and 10mm in case of accessible stenosis with balloon enteroscopy)
* Dilated stenosis according to endoscopist criteria (pass or no the endoscopy)
* Patient capable of participate in the examinations required by the study
* Patient after being informed, give his/her informed consent in writing

Exclusion Criteria:

* Patients with large intestinal stenosis (more than 6cm) and multiples
* Patients with previous or actual treatment with anti-tumor necrosis factor (anti-TNF) drugs
* Patients with positive serology to hepatitis B virus(HBV),hepatitis C virus (HCV), or HIV
* Patients with positive screening to Tuberculosis(positive PPD)
* Established contraindication to anti-TNF drugs
* Existence of fistulous tracts associated with intestinal stenosis
* Neoplastic process associated with stenosis or in another location
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02-14; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Success of endoscopic dilatation | at week 8
  Successful dilatation means the passage of the endoscope (or enteroscopy colonoscope) through the stenosis

SECONDARY OUTCOMES:
Stenosis measure | baseline
  The endoscopic stenosis diameter will be estimated pre and post-dilatation
success of endoscopic dilatation | at week 52
  The success of endoscopic dilatation at week 52 means absence of clinical subocclusion, no necessity of surgical nor endoscopic dilatation
Mucosal healing | at week 8
  * Anastomotic strictures: We define mucosal healing as a Rutgeerts < or equal 2 with at least 1 point of improvement (añadir el score)
  * Primary strictures: Absence of ulcers after treatment
Histological cure | at week 8
  We consider histological cure if:
  * Epithelial damage is < or equal 1
  * Architectural changes is < or equal 1
  * Infiltration of mononuclear cells in lamina propria is < or equal 1
  * Polymorphonuclear cells in the lamina propria = 0
  * Polymorphonuclear cells in epithelium = 0
  * Absence of erosions and ulcers (based ib scoring system for Histologic Abnormalities in Crohn's disease Mucosal Biopsy Specimens - Title: Early lesions of recurrent Crohn's disease caused by infusion of intestinal contents in excluded ileum Author(s): D'Haens, Geert R.; Geboes, Karel; Peeters, Mark; et al. Source: Gastroenterology Volume: 114 Issue: 2 Pages: 262-267 Published: Feb., 1998)
proportion of patients that develop anti-adalimumab antibodies | at the end of the study
adverse events | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Begoña González Suarez, MD, Principal Investigator — Hospital Clinic of Barcelona; Lucía Márquez, MD, Principal Investigator — Hospital del Mar; Alfredo Mata, MD, Principal Investigator — Hospital de Sant Joan Despí Moisès Broggi; Carlos Huertas, MD, Principal Investigator — Hospital Josep Trueta; Lidia Argüello, MD, Principal Investigator — Hospital La Fe; Cecilia González, MD, Principal Investigator — Gregorio Marañón Hospital; Ana Echarri, MD, Principal Investigator — Complexo Hospitalario Arquitecto Marcide-Novoa Santos; Carme Loras, Principal Investigator — Hospital Mútua Terrassa; Maria D Martín Arranz, Principal Investigator — Hospital Universitario La Paz; Manuel Barreiro, Principal Investigator — Complexo Hospitalario de Santiago; Yago González, Principal Investigator — Hospital Universitario Puerta del Hierro; Beatriz Sicília, Principal Investigator — Complejo asistencial Universitario de Burgos; Sam Korrhami, Principal Investigator — Hospital Son Espases; Ana Gutiérrez, Principal Investigator — Hospital General Universitario de Alicante
Locations (13):
- Spain (13):
  - Complexo Hospitalario Arquitecto Marcide -Novoa Santos, Ferrol, A Coruña
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Puerta del Hierro, Majadahonda, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Complejo asistencial universitario de Burgos, Burgos
  - Hospital Josep Trueta, Girona
  - Hospital La Paz, Madrid
  - Hospital La Fe, Valencia